CLINICAL TRIAL: NCT02524574
Title: Tomography Positron Emission Assessment of the Impact of Cardiac Rehabilitation on Coronary Endothelial Function in Cardiac Failure
Acronym: TEP-READ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-089
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Rehabilitation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cardiac Rehabilitation (Experimental)
  Interventions: Procedure: cardiac Rehabilitation; Other: Tomography Positron Emission

INTERVENTIONS:
Procedure: cardiac Rehabilitation
Other: Tomography Positron Emission

SUMMARY:
In patients with heart failure, the drive to the effort has demonstrated its safety and its interest. Patients with heart failure, endothelium-dependent peripheral vasodilatation is impaired by decreased activity of endothelial NO synthase. The rehabilitation training significantly improves peripheral endothelial function, and this improvement is correlated to the increase in exercise capacity. The impact on coronary endothelial function remains poorly documented, especially in non-ischemic dilated heart disease.

The main objective of this study is to investigate the effectiveness of cardiac rehabilitation on the restoration of coronary endothelial function in cardiac failure patient evaluated with Tomography Positron Emission 15O-H2O.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure with nonischemic dilated cardiomyopathy
* Class II-III NYHA (New York Heart Association)
* Having no contra-indication to the effort
* Fraction Ejection ≤ 40%
* patient who will have cardiac rehabilitation
* Age over 18 years
* informed consent signed
* patient with a social security scheme

Exclusion Criteria:

* Hypertension> 160/90 mmHg
* High cholesterol level > 6.0 mmol / l
* Diabetes known and treated
* Active smoking
* Valvular heart disease, congenital or ischemic
* Pregnant or breastfeeding women
* Age <18 years
* Major Adult guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Rate of myocardial blood flow during the cold test | change over baseline and after 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Cardiologie, Caen, France

REFERENCES:
- [Result] Legallois D, Belin A, Nesterov SV, Milliez P, Parienti JJ, Knuuti J, Abbas A, Tirel O, Agostini D, Manrique A. Cardiac rehabilitation improves coronary endothelial function in patients with heart failure due to dilated cardiomyopathy: A positron emission tomography study. Eur J Prev Cardiol. 2016 Jan;23(2):129-36. doi: 10.1177/2047487314565739. Epub 2014 Dec 18. PMID 25525058
- [Result] Tuffier S, Legallois D, Belin A, Joubert M, Bailliez A, Redonnet M, Agostini D, Manrique A. Assessment of endothelial function and myocardial flow reserve using (15)O-water PET without attenuation correction. Eur J Nucl Med Mol Imaging. 2016 Feb;43(2):288-295. doi: 10.1007/s00259-015-3163-x. Epub 2015 Aug 18. PMID 26280980